CLINICAL TRIAL: NCT06813755
Title: Effect of Ultrasound (USG)-Guided Pericapsular Nerve Group (PENG) Block on Pain During Participant Positioning for Spinal Anesthesia in Hip Fracture Surgery: a Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group (PENG) Block on Pain During Participant Positioning for Spinal Anesthesia in Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Gul Cakmak, medical doctor, Marmara University
Other Study IDs: E-10840098-202.3.02-6997
Record Dates: First submitted 2024-12-09; First posted 2025-02-07 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Femur Fracture; Hip Surgery
Keywords: peng block; regional anesthesia; geriatric population
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Procedure: PENG Block Pericapsular Nerve Group Block: Active Comparator: PENG Block For patients with hip fracture and having hip surgery this study evaluates the analgesic effects of Pericapsular Nerve Group (PENG) block for positioning before spinal anesthesia.
- Drug: Conventional intravenous sedoanalgesia (ketamine) standardised intravenous sedoanalgesia agent: Active Comparator: Control in this group, standardised sedoanalgesia doses (drug: ketamine) will be used for analgesia for positioning pain

SUMMARY:
Hip fracture surgery is a common orthopedic procedure, especially in elderly patients. These fractures are quite common in adults over the age of 65, and the one-year mortality rate ranges from 12% to 37%. Recent studies have suggested that general anesthesia and spinal anesthesia are not superior to each other in patients undergoing hip fracture surgery. Untreated/poorly managed perioperative pain is directly linked to delirium, poor prognosis, and secondary chronic pain in hip fracture patients. Therefore, considering the associated mortality, morbidity, and early recovery, control of perioperative pain should be one of the highest priorities of the anesthesiologist, regardless of the anesthesia method used.

DETAILED DESCRIPTION:
Ultrasonography (USG)-guided regional anesthesia techniques are often used as part of multimodal analgesia in the management of perioperative pain in patients with hip fractures. One of the most recently described blocks used in hip fracture surgery, the USG-guided pericapsular nerve group (PENG) block, aims to directly block the articular branch of the femoral nerve, the articular branch of the obturator nerve, and the accessory obturator nerve, which selectively innervates the anterior aspect of the hip capsule. Case reports and a limited number of clinical studies have reported that PENG block is effective in managing acute fracture-related pain, neuraxial anesthesia positioning pain, and postoperative pain in hip fracture patients.

In this study, investigators aimed to investigate the effect of USG-guided PENG block on positional pain before spinal anesthesia in patients undergoing surgery for hip fractures and to compare this effect with intravenous ketamine.

In addition, investigators aimed to investigate the effect of PENG block on pain scores, perioperative opioid consumption, time to first analgesic requirement in the postoperative period, and quality of recovery in the first 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

hip fracture aged between 35 and 90 years old

Exclusion Criteria:

contraindications for spinal anesthesia and PENG block impaired cognition or dementia multiple fractures any previous analgesic administration during the last 12 hours

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 participants older than the age of 40 who will undergo hip fracture surgery under spinal anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Pain scores on the Numeric Rating Scale (NRS) | Group A: 5 minutes after intervention (intravenous opioid), Group B: 20 minutes after intervention (PENG block)
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Duration of spinal anesthesia performance | Group A: 5 minutes after intervention (intravenous ketamine), Group B: 20 minutes after intervention (PENG block)
  It will be measured in "minutes", from the start of positioning maneuvers to the spinal needle removal
Quality of patient's position | Group A: 5 minutes after intervention (intravenous ketamine), Group B: 20 minutes after intervention (PENG block)
  The position will be characterized as "unsatisfactory", "satisfactory", "good" or "very good"
Analgesic consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a rescue analgesia agent (tramadol).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aygun H, Tulgar S, Yigit Y, Tasdemir A, Kurt C, Genc C, Bilgin S, Senoglu N, Koksal E. Effect of ultrasound-guided pericapsular nerve group (PENG) block on pain during patient positioning for central nervous blockade in hip surgery: a randomized controlled trial. BMC Anesthesiol. 2023 Sep 15;23(1):316. doi: 10.1186/s12871-023-02245-3. PMID 37715173